CLINICAL TRIAL: NCT04774445
Title: Effectiveness of MyCancerGene to Optimize Genetic Testing Outcomes
Acronym: MyCancerGene
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC 10919; 832628 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Genetic Predisposition
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individuals randomized to this arm will receive immediate access to the Interactive Health Communication Application.
  Interventions: Behavioral: MyCancerGene
- Usual Care Group (No Intervention): Individuals randomized to this arm will receive the standard clinical practice.

INTERVENTIONS:
Behavioral: MyCancerGene — Interactive Health Communication Application
  Arms: Intervention Group

SUMMARY:
This protocol aims to evaluate the efficacy of a theoretically and stakeholder informed patient-centered genetic Interactive Health Communication Application to increase patient understanding of, and affective and behavioral responses to genetic testing. The study investigators hypothesize that the intervention will be associated with increases in knowledge, decreases in distress, increases in communication with relatives and health care providers, and increases in performance of risk reducing health behaviors.

DETAILED DESCRIPTION:
As clinical practice increasingly use multi-gene testing, many patients are left with unknowns after genetic testing. Many have results that are unclear and may or may not be associated with any risk for cancer (Variants of Uncertain Significance), or mutations in genes with very limited information about disease risk or the best medical management. Importantly, many of these uncertainties will be clarified over time, but there is a need for effective ways of communicating these updates to patients who had testing months or years ago. In some cases, there may be multiple updates over time. To address this, this study will provide patients access, using an Interactive Health Communication Application, MyCancerGene, to information about their genetic testing, their specific results and the implications, the ability to print reports and other materials for their relatives and other health care providers and to assess if there has been a change in the personal or family history. Additionally, patients can contact their genetic provider through MyCancerGene and the cancer genetics team can send out updates to patients about their individual results or about new information about risk estimates or screening recommendations. The study investigators hypothesize that MyCancerGene will be associated with increases in knowledge, decreases in distress, increases in communication with relatives and health care providers, and increases in cancer screening and risk reducing health behaviors. After 12 months, all patients will have access to MyCancerGene, which will aid in understanding who benefits most and least from this intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English Speaking
* Male or Female
* Internet and/or mobile access
* Previously received clinical genetic counseling and testing for hereditary cancer syndromes (up to 60 days prior to recruitment)

Exclusion Criteria:

•No internet and/or mobile access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The KnowGene Scale | Baseline - 18 Months
  Change in Knowledge. Score Range = 0-16. Higher score = Better outcome
Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline - 18 Months
  Change in General Anxiety and Depression. Score Range = 4-20 for Anxiety/4-20 for Depression. Lower score = Better outcome

SECONDARY OUTCOMES:
Multi-dimensional Impact of Cancer Risk Assessment Questionnaire (MICRA) | Baseline - 18 Months
  Change in Uncertainty. Score Range = 0-85. Lower score = Better outcome
Impact of Events Scale (IES) | Baseline - 18 months
  Change in Disease-Specific Distress. Score Range =0-40. Lower score = Better outcome
Test Result Recall | Baseline - 18 months
  Single item assessing participants' ability to accurately recall their genetic test result. Single answer multiple choice: Positive, Negative, Variant of Uncertain Significance
Perceptions of Genetic Disease | Baseline - 18 months
  Quantitative scales assessing changes in perceived risk, timeline and utility.
Behavioral Risk Factor Surveillance System Questionnaire (BRFSS) | Baseline - 18 months
  Changes in modifiable cancer lifestyle behaviors. Yes/No responses.
Health and Diet Survey Dietary Guidelines Supplement | Baseline - 18 months
  Changes in diet and exercise. Yes/No responses.
Sharing Genomic Information with Relatives (adapted from the PHENX Toolkit) | Baseline - 18 months
  Assesses the number of relatives and health care providers patients share genetic test results with

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Bradbury, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States